CLINICAL TRIAL: NCT03438058
Title: Complement-activating Anti-human Leucocyte Antigen Donor Specific Antibodies in Solid Organ Transplantation: A Systematic Review and Meta-analysis
Brief Title: Complement-activating Anti-human Leucocyte Antigen Donor Specific Antibodies in Solid Organ Transplantation
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Principal Investigator, Professor Alexandre Loupy, Professor Alexandre Loupy, Paris Translational Research Center for Organ Transplantation
Other Study IDs: ALPINIST001
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Organ Transplant Recipients
Keywords: Solid Organ Transplantation; Graft survival; Rejection; Complement-activating anti-HLA DSA; Meta-analysis; Prognosis
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- With complement-activating anti-HLA DSAs: Patients with complement-activating anti-HLA DSAs either C1q, C3d, C4d and IgG subclass
  Interventions: Other: Graft survival and/or Rejection appearance
- Without complement-activating anti-HLA DSAs: Patients with anti-HLA DSAs but without the ability to activate the complement (either C1q, C3d, C4d and IgG subclass)
  Interventions: Other: Graft survival and/or Rejection appearance
- Without DSAs and without complement-activating DSAs: Matching group of patients without DSAs and without complement-activating DSAs
  Interventions: Other: Graft survival and/or Rejection appearance

INTERVENTIONS:
Other: Graft survival and/or Rejection appearance

SUMMARY:
This project will involve a systematic literature review and meta-analysis of studies assessing the impact of complement-activating anti-Human Leukocyte Antigen (HLA) donor specific antibodies (DSA) on the allograft survival rate and on the rejection rate.

This meta-analysis will assess the role of complement activating anti-HLA DSAs across the entire transplant field including kidney, liver, lung and heart transplant recipient's studies.

DETAILED DESCRIPTION:
BACKGROUND:

Organ transplantation has emerged as the treatment of choice for patients with end-stage chronic disease, which is an increasing burden in industrialized and newly-industrializing societies. For example, the global burden of end-stage renal disease in 2017 is estimated to be 3,900,000 with an ~6% growth rate, which is significantly greater than world population growth. Today, over one million people worldwide live with organ transplants, and another 120,000 organs transplanted each year.

Despite progress in transplantation, allograft rejection remains a major threat to allograft health, with thousands of allografts failing every year worldwide due to organ rejection. Failed allografts create immediate and severe consequences for patients in terms of mortality and morbidity, while generating billions in extra costs to health care systems.

One of the most important advances in transplant medicine was the recognition that anti-human lymphocyte antigen (anti-HLA) antibodies are destructive. Recently, lots of studies recognized the capacity of anti-HLA antibodies to activate complement and determined that complement activation magnifies the cytotoxic potential of these antibodies. Over the last decade, studies have reported that complement-activation is highly associated with allograft rejection and failure, with varying magnitudes of effect. In addition, more recent studies have suggested that beyond kidney allografts, these antibodies could have a broad universal deleterious effect in other solid organ transplants such a heart, liver and lung allografts.

MAIN OUTCOMES AND MEASURES:

Evaluate the clinical relevance of complement-activating anti-HLA antibodies at a population level, by performing a meta-analysis across solid organ transplants (kidney, liver, heart and lung transplant patients) to determine the magnitude of the association between the presence of complement-activating antibody and the related risk for allograft failure and risk of rejection.

DESIGN:

This meta-analysis will report in adherence with the preferred reporting items for systematic reviews and meta-analyses (PRISMA) and the reporting Meta-Analyses of Observational Studies in Epidemiology (MOOSE).

A comprehensive search will be design and conduct by an experienced librarian with input from the study investigators. Controlled vocabulary supplemented with keywords will be used to search for complement-activating anti-human leucocyte antigen donor-specific antibodies in human solid organ transplantation in any language. The following databases will be included: Ovid MEDLINE In-Process & Other Non-Indexed Citations, Ovid MEDLINE, Ovid EMBASE, Ovid Cochrane Central Register of Controlled Trials, Ovid Cochrane Database of Systematic Reviews, and Scopus.

ELIGIBILITY:
Inclusion Criteria:

* Study design:

Studies of any relevant design and in any language on the impact of complement-activating anti-HLA DSAs on long-term graft survival and/or the risk of rejection will be initially selected.

* eligible studies: The eligible studies include all solid organ transplant patients (kidney, liver, lung, heart, and intestinal transplantation), both adult or paediatric patients.
* Measurement:

Anti-HLA DSAs detect by the single antigen Luminex bead technique (SAB) will be required for the DSA detection technique. Complement-activating anti-HLA DSAs will be defined according to their ability to bind C1q, C3d, and C4d or their IgG3 subclass.

Exclusion Criteria:

* Animal studies
* Ex vivo studies
* Methodological studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible studies include all solid organ transplant patients (kidney, liver, lung, heart, and intestinal transplantation), both adult or paediatric patients in which complement-activating anti-HLA DSAs have been measured (either C1q, C3d, and C4d or their IgG3 subclass). In those studies data on allograft survival and rejection rate have to be measure.
Sampling Method: Non-Probability Sample
Enrollment: 7547 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Allograft Survival rate | death censored allograft survival at minimum 1 year of follow up
  To assess the impact of complement-activating anti-Human Leukocyte Antigen (HLA) donor specific antibodies (DSA) on the allograft survival rate in solid organ transplant patients (Heart, Kidney, Lung, Liver and Small Bowel transplant recipients)

SECONDARY OUTCOMES:
Allograft Rejection rate | rejection rate during follow up (at minimum 3 months post transplantation) or rejection defined by biopsy at inclusion
  To evaluate the impact of complement-activating anti-HLA DSA on the risk of antibody mediated rejection or biopsy proven histological allograft injury

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lefaucheur, PhD, Principal Investigator — Paris Translational Research Center for Organ Transplantation; Alexandre Loupy, PhD, Principal Investigator — Paris Translational Research Center for Organ Transplantation

IPD SHARING:
Plan to Share IPD: No
No access to the individual participant data

REFERENCES:
- [Derived] Bouquegneau A, Loheac C, Aubert O, Bouatou Y, Viglietti D, Empana JP, Ulloa C, Murad MH, Legendre C, Glotz D, Jackson AM, Zeevi A, Schaub S, Taupin JL, Reed EF, Friedewald JJ, Tyan DB, Susal C, Shapiro R, Woodle ES, Hidalgo LG, O'Leary J, Montgomery RA, Kobashigawa J, Jouven X, Jabre P, Lefaucheur C, Loupy A. Complement-activating donor-specific anti-HLA antibodies and solid organ transplant survival: A systematic review and meta-analysis. PLoS Med. 2018 May 25;15(5):e1002572. doi: 10.1371/journal.pmed.1002572. eCollection 2018 May. PMID 29799874